CLINICAL TRIAL: NCT00558077
Title: Laparoscopic Ovarian Diathermy or Metformin Plus Clomiphene Citrate Administration as Second-Line Treatment for Infertile Anovulatory Patients With Polycystic Ovary Syndrome: a Randomized Controlled Trial
Brief Title: Second-Line Treatments for Anovulatory Infertility in PCOS Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Magna Graecia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01/2003
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Last update posted 2007-11-14 (Estimated); Status verified 2007-11

CONDITIONS: Polycystic Ovary Syndrome; Infertility; Anovulation
Keywords: Anovulation; Clomiphene citrate; Fertility; Metformin; Ovulation induction; PCOS; Sterility; Treatment; Clomiphene citrate-resistance
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility; Anovulation | interventions — Metformin; Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Metformin plus clomiphene citrate
  Interventions: Drug: Metformin plus clomiphene citrate
- B (Active Comparator): Laparoscopic ovarian drilling
  Interventions: Procedure: Laparoscopic ovarian drilling

INTERVENTIONS:
Drug: Metformin plus clomiphene citrate — Metformin administration will start from 3rd day of a P-induced withdrawal bleeding with a dose of 850 mg (1 tablet daily) and increasing the dosage after one week up to 1700 mg/day (two tablets daily). Clomiphene citrate CC will be administered for five days beginning on cycle day 3rd of a P-induced withdrawal bleeding using a starting dose of 50 mg daily. If ovulation will not occur, the dose will be increased by 50 mg in successive cycles until the ovulation will be achieved or up to a maximal dose of 150 mg daily.
  Arms: A
Procedure: Laparoscopic ovarian drilling — Laparoscopic ovarian drilling will be performed as follows: according to ovary size three to six punctures will be performed at each ovary inserting an insulated needle cautery of 36 mm perpendicularly as possible to the ovarian surface with a cutting current of 100 watt power. Then, the needle will be activated for 2-3 seconds at each point using a coagulating current of 40 watt power. At completion of the procedure, the ovarian surface will be washed with a crystalloid solution and all injured areas will be completely covered with hyaluronic acid gel.
  Arms: B

SUMMARY:
To date, it is still unclear the potential role of laparoscopic ovarian diathermy (LOD) in the management of polycystic ovary syndrome (PCOS)-related anovulatory infertility. Metformin administration, alone or combined with clomiphene citrate (CC), has shown to be an effective and attractive second-line treatment for ovulation induction in women with polycystic ovary syndrome (PCOS) after failure of CC treatment. The aim of the present study will be to compare in a randomized controlled fashion the efficacy of LOD with metformin plus CC administration in the treatment of the CC-resistant PCOS patients.

DETAILED DESCRIPTION:
A total of 50 primary infertile anovulatory PCOS patients with documented CC-resistance will be enrolled and randomized into two groups of treatment of 25 subjects each. Group A will undergo diagnostic laparoscopy followed by metformin plus CC, whereas group B will undergo LOD followed by observation. Anovulatory patients will receive IM progesterone. The treatment will be of six months followed by nine-month of observation for pregnant patients. The incidence of spontaneous menses, and the pregnancy, abortion, and live-birth rates will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* PCOS
* Clomiphene citrate-resistance
* Anovulation
* Infertility

Exclusion Criteria:

* Age < 18 or > 35 years
* Body mass index >35
* Neoplastic, metabolic, endocrine, hepatic, renal, and cardiovascular disorders or other concurrent medical illnesses
* Current or previous use of oral contraceptives, glucocorticoids, antiandrogens, ovulation induction agents, antidiabetic and anti-obesity drugs or other drugs affecting hormone levels, carbohydrate metabolism, or appetite
* Pelvic diseases
* Previous pelvic surgery
* Suspected peritoneal factor infertility/subfertility
* Tubal or male factor infertility or sub-fertility

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2003-02; Study Completion 2005-10

PRIMARY OUTCOMES:
Live-birth rate | fifteen months

SECONDARY OUTCOMES:
Spontaneous menses | six months
Pregnancy rate | six months
Abortion rate | fifteen months

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Palomba, MD, Principal Investigator — Department of Obstetrics and Gynecology, University "Magna Graecia" of Catanzaro; Fulvio Zullo, MD, Study Chair — Department of Obstetrics and Gynecology, University "Magna Graecia" of Catanzaro
Locations (1):
- "Pugliese" Hospital, Catanzaro, Catanzaro/Italy, Italy

REFERENCES:
- [Background] Palomba S, Orio F Jr, Falbo A, Manguso F, Russo T, Cascella T, Tolino A, Carmina E, Colao A, Zullo F. Prospective parallel randomized, double-blind, double-dummy controlled clinical trial comparing clomiphene citrate and metformin as the first-line treatment for ovulation induction in nonobese anovulatory women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2005 Jul;90(7):4068-74. doi: 10.1210/jc.2005-0110. Epub 2005 Apr 19. PMID 15840746
- [Background] Palomba S, Orio F Jr, Nardo LG, Falbo A, Russo T, Corea D, Doldo P, Lombardi G, Tolino A, Colao A, Zullo F. Metformin administration versus laparoscopic ovarian diathermy in clomiphene citrate-resistant women with polycystic ovary syndrome: a prospective parallel randomized double-blind placebo-controlled trial. J Clin Endocrinol Metab. 2004 Oct;89(10):4801-9. doi: 10.1210/jc.2004-0689. PMID 15472166